CLINICAL TRIAL: NCT06398925
Title: A Phase I, First-in-human, Randomised, Double-blind, Placebo-controlled, Single Ascending Oral Dose, Safety, Tolerability and Pharmacokinetic Study to Investigate the Effects of OCT461201 in Healthy Volunteers
Brief Title: Single Ascending Oral Dose Study to Investigate the Effects of OCT461201 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford Cannabinoid Technologies Holdings PLC (Industry)
Collaborators: Simbec-Orion Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCT-001-2023
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Phase 1; Single Ascending Dose; Health volunteer

STUDY DESIGN:
Intervention Model Description: Single ascending dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, randomised study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- OCT461201 Dose Level 1 (Experimental): Single ascending dose of OCT461201 10 mg
  Interventions: Drug: OCT461201 50 mg; Drug: Placebo
- OCT461201 Dose Level 2 (Experimental): Single ascending dose of OCT461201 50 mg
  Interventions: Drug: OCT461201 100 mg; Drug: Placebo
- OCT461201 Dose Level 3 (Experimental): Single ascending dose of OCT461201 150 mg
  Interventions: Drug: OCT461201 150 mg; Drug: Placebo
- OCT461201 Dose Level 4 (Experimental): Single ascending dose of OCT461201 450 mg
  Interventions: Drug: OCT461201 450 mg; Drug: Placebo
- Placebo (Placebo Comparator): Single dose of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OCT461201 50 mg — Oral capsule
  Arms: OCT461201 Dose Level 1
Drug: OCT461201 100 mg — Oral capsule
  Arms: OCT461201 Dose Level 2
Drug: OCT461201 150 mg — Oral capsule
  Arms: OCT461201 Dose Level 3
Drug: OCT461201 450 mg — Oral capsule
  Arms: OCT461201 Dose Level 4
Drug: Placebo — Placebo capsule

SUMMARY:
A study in healthy volunteers to evaluate the safety, tolerability and pharmacokinetics of OCT461201. The study included a screening period, a single dose of study treatment or placebo and a follow up period.

DETAILED DESCRIPTION:
A phase 1, randomised, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of OCT461201 in healthy participants following ascending single doses.

The study comprised a screening period (Day -35 to Day -2), a treatment period (Day -1 to Day 3) and a post-study follow-up visit 4 - 8 days following administration of OCT461201 or placebo (i.e., Day 5 - 9). A dose leader design was implemented with 2 participants being dosed on the first dosing day (1 randomised to placebo, 1 to active drug) and the remainder of the cohort dosed at least 24 hours later pending an acceptable safety profile in the dose leader group. Safety and Pharmacokinetic data was reviewed by the Dose Escalation Review Committee before escalation to the next cohort/dose level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participant, between 15 and 55 years of age inclusive at screening
* Body mass index (BMI) of 18-30 kg/m2
* No clinically significant history of previous allergy/sensitivity to compounds similar to experimental drug or any of its excipients
* No clinically significant results for serum biochemistry, haematology and/or urine analysis within 35 days before first dose of Investigational Medicinal Product (IMP)
* No clinically significant abnormalities in 12-lead ECG within 35 days before dose of IMP
* Available to complete the study including all follow up visits

Exclusion Criteria:

* Clinically significant history of gastrointestinal disorder likely to influence IMP absorption
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction
* Participation in a new chemical entity clinical study within the previous 3 months or 5 half-lives, whichever was longer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events during the study assessed as mild, moderate or severe | Day 1-9

SECONDARY OUTCOMES:
Pharmacokinetic parameter: Cmax | Day 1-3
  Maximum observed concentration
Pharmacokinetic parameter: AUC | Day 1-3
  Overall exposure
Pharmacokinetic parameter: t1/2 | Day 1-3
  Terminal elimination half life

CONTACTS AND LOCATIONS:
Locations (1):
- Simbec-Orion, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No